CLINICAL TRIAL: NCT03065101
Title: Functional Advantages of TRIGEN™ INTERTAN™ Over Sliding Hip Screw in Subjects With Trochanteric Hip Fracture: A Randomised Controlled Trial
Brief Title: Trigen InterTAN vs Sliding Hip Screw RCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Smith & Nephew Orthopaedics AG (Industry)
Responsible Party: Sponsor
Organization: Smith & Nephew, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-3031-01
Record Dates: First submitted 2016-03-24; First posted 2017-02-27 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trigen Intertan (Other): * Unique integrated interlocking screw and trapezoidal nail shape
  * Resistance to femoral head rotation and cut-out
  * Active compression through linear motion without rotation
  * Single subtrochanteric lag screw option for stable fractures below lesser trochanter
  * Preloaded cannulated set screw converts construct to fixed angle device
  * Small proximal diameter of the nail promotes preservation of the lateral wall of the greater trochanter and gluteus medius tendon
  * Clothespin tip for stress modulation in femoral shaft
  * Potential for improved patient mobility and recovery
  Manufactured by Smith & Nephew Inc., 1450 Brooks Road, Memphis, TN 38116, U.S.A.
  Interventions:
  Randomisation to either Trigen Intertan or Sliding Hip Screw, Post-Surgery Follow Up
  Interventions: Device: Trigen Intertan; Other: Post-Surgery Follow Up
- Sliding Hip Screw (Other): SHS is a generic term for a group of devices used for internal fixation of trochanteric hip fractures. Also known as Compression Hip Screw or Dynamic Hip Screw. All devices feature a lag screw inserted into the femoral neck and a side plate held in place by cortical screws inserted into the proximal femoral shaft.
  Therapeutic effect is achieved by guided collapse, where the lag screw can slide in the barrel of the side plate which compresses the fracture as the patient begins to weight-bear.
  Participating sites may use whichever brand of SHS is currently in use.
  Interventions:
  Randomisation to either Trigen Intertan or Sliding Hip Screw, Post-Surgery Follow Up
  Interventions: Other: Post-Surgery Follow Up; Device: Sliding Hip Screw

INTERVENTIONS:
Device: Trigen Intertan — While both the Trigen InterTAN and Sliding Hip Screw are marketed and demonstrated to be suitable for treatment of the study indication, the randomisation is considered an intervention as it may be contrary to the treatment chosen by the surgeon were the patient not a study subject.
  Arms: Trigen Intertan
Other: Post-Surgery Follow Up — The current clinical trend is for minimal follow up post-surgery, unless indicated by complications. The study protocol indicated that follow up telephone visits are to be performed at 8 weeks, 12 weeks and 12 months post-surgery and an outpatient follow up visit at 6 months post-surgery. While most outcome measures are conducted via questionnaire, the increase in follow up means that subjects may be exposed to increased ionising radiation.
Device: Sliding Hip Screw — Sliding Hip Screw
  Arms: Sliding Hip Screw

SUMMARY:
The purpose of this study is to compare the Trigen InterTAN Intramedullary nail to Sliding Hip Screws in AO/OTA 31-A1 and A2 intertrochanteric hip fractures.

DETAILED DESCRIPTION:
A multicentre, randomised controlled trial, conducted in the UK will recruit 180 subjects, randomised to receive either the Trigen InterTAN Nail or the Sliding Hip Screw.

Subjects presenting at participating hospitals with AO/OTA 31-A1 or A2 fractures will be assessed against the eligibility criteria and approached for Informed Consent.

Subjects who are considered eligible and who have provided Informed Consent will be randomised using iDataFax to one of the two treatment options.

Subjects will be operated on according to standard procedure and the Instructions for Use.

A daily inpatient assessment will record the subjects use of opioid pain medication.

Subjects will be assessed at the time of discharge to record their residential and ambulatory status, Functional Independence Measure, Get Up and Go Test and opioid usage.

At 8 weeks and 12 weeks post surgery, subjects will be contacted by telephone to confirm their residential and ambulatory status, Functional Independence Measure, modified Harris Hip Score and Euroqol-5D.

At 6 months post surgery, subjects will attend an outpatient visit to have a follow up radiograph, Get Up and Go Test, residential and ambulatory status, Functional Independence Measure, modified Harris Hip Score and Euroqol-5D.

At 12 months post surgery, subjects will be contacted by telephone to confirm their residential and ambulatory status, Functional Independence Measure, modified Harris Hip Score and Euroqol-5D.

Adverse events, device deficiencies and reoperations will be recorded as and when they occur throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* has closed trochanteric hip fracture (AO/OTA 31-A1 or A2) requiring treatment with internal fixation
* has injury due to low energy trauma
* is independently ambulatory in living environment prior to injury (walking aids permitted)
* is >60 years of age
* is willing and able to participate in required follow-up visits at the investigational site and to complete study procedures and questionnaires
* has consented to participate in the study by signing the Ethics Committee (EC) approved ICF
* has definitive fracture fixation <72h from admission

Exclusion Criteria:

* has any additional injury or disability affecting mobility or affecting use of walking aids
* has a pathological fracture (excluding osteoporotic fracture)
* has an existing implant in study hip
* has diagnosis of an immunosuppressive disorder
* has an active infection, treated or untreated, systemic or at the site of the - has a condition that may interfere with the outcome of the study, including but not limited to: Paget's disease, Charcot's disease, vascular insufficiency, muscular atrophy, uncontrolled diabetes, renal insufficiency or neuromuscular disease
* has a BMI >40
* has an inadequate bone stock to support the device which would make the procedure unjustifiable, including but not limited to: severe osteopenia/osteoporosis or family history of severe osteoporosis/osteopenia
* is pregnant or plans to become pregnant during the course of the study
* is a prisoner or is facing impending incarceration
* in the opinion of the PI, has an emotional or neurological condition that would interfere with their ability or willingness to participate in the study including mental illness, mental retardation, and drug or alcohol abuse
* is entered in another investigational drug, biologic, or device study or has been treated with an investigational product in the past 30 days
* is known to be at risk for lost to follow-up, or failure to return for scheduled visits

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Functional Independence Measure (motor portion) | 8 weeks post-surgery
  The FIM instrument is a basic indicator of severity of disability. Comprises 18 items assessed against a seven point ordinal scale, where the higher the score for an item, the more independently the patient is able to perform the tasks assessed by that item. Total scores range from 18 to 126. The items are divided into 13 Motor items and 5 Cognitive Items. The rating scale designates major graduations in behaviour from dependence to independence. The scale provides for the classification of individuals by their ability to carry out an activity independently, versus their need for assistance from another person or a device. If help is needed the scale assesses the degree of that need.
  Patient reported outcome.

SECONDARY OUTCOMES:
Functional Independence Measure | 12 weeks, 6 months and 12 months post-surgery
  The FIM instrument is a basic indicator of severity of disability. Comprises 18 items assessed against a seven point ordinal scale, where the higher the score for an item, the more independently the patient is able to perform the tasks assessed by that item. Total scores range from 18 to 126. The items are divided into 13 Motor items and 5 Cognitive Items. The rating scale designates major graduations in behaviour from dependence to independence. The scale provides for the classification of individuals by their ability to carry out an activity independently, versus their need for assistance from another person or a device. If help is needed the scale assesses the degree of that need.
  Patient reported outcome.
Get Up and Go Test | Discharge (estimated 2 weeks post-surgery) and 6 months post-surgery
  Requires the study subject to;
  1. Sit comfortably in a straight-backed chair
  2. Rise from the chair
  3. Stand still momentarily
  4. Walk a short distance (approximately 3 metres)
  5. Turn around
  6. Walk back to the chair
  7. Turn around
  8. Sit down in the chair Movements are observed for any deviation from a confident, normal performance and recorded as;
  1. Normal 2. Very slightly abnormal 3. Mildly abnormal 4. Moderately abnormal 5. Severely abnormal Subjects will be scored as above and whether any mobility aids were required. The GUG Test will be supervised and recorded by study staff.
Residential Status Questionnaire | Pre-Op (Day prior to or day of surgery), Discharge (estimated 2 weeks post-surgery), 8 weeks, 12 weeks, 6 months and 12 months post-surgery
  Pre-operatively it will be recorded what the subjects' residential status was prior to injury, whether they were;
  * living at home independently
  * living at home with additional care
  * living in sheltered housing
  * living in a care institution At discharge and thereafter it will be recorded which of these living environments the subject is discharged to with the additional option of;
  * NHS rehabilitation
Ambulatory Status Questionnaire | Pre-Op (Day prior to or day of surgery), Discharge (estimated 2 weeks post-surgery), 8 weeks, 12 weeks, 6 months and 12 months post-surgery
  Pre-operatively it will be recorded what the subjects' ambulatory status was prior to injury inside and outside their living environment, whether they were;
  * Walking unaided
  * Walking with aids
    * 1 stick
    * 2 sticks
    * Frame
    * Wheelchair (Note: Wheelchair use inside the living environment pre-operatively is an exclusion criterion. Wheelchair use outside the living environment is permitted if the subject is walking unaided or with stick(s) or frame inside the home) Ambulatory status will be recorded at discharge and at all Follow-Up timepoints thereafter.
Radiographic Assessment (calculation of medialisation, shortening and tip-apex distance) | Pre-Op (Day prior to or day of surgery), immediately post-op and 6 months post-surgery
  A pre-operative low centred anteroposterior (AP) pelvis and lateral hip X-ray radiograph will be taken for diagnostic purposes. If a deformity is noted, a full length AP and lateral femur X-ray will be conducted in addition.
  The post-operative low centre AP pelvis and lateral hip X-ray radiographic assessment will record;
  * femoral shortening
  * femoral shaft medialisation
  * offset
  * tip-apex distance If a long nail is used or if there are concerns over fixation, a full length AP and lateral femur X-ray will be conducted in addition.
Modified Harris Hip Score | 8 weeks, 12 weeks, 6 months and 12 months post-surgery
  The HHS was developed to assess the results of hip surgery, first described in 1969 . A modified version (mHHS) is used in this study which records the subjects' experience of pain (worth a maximum of 44 points) and activities of daily living and gait (worth a maximum of 47 points). A higher score is associated with a better outcome. Questions include pain experienced, the distance the subject can walk, ability to put on socks and shoes, ability to use public transportation, supports needed, limp, ability to use stairs and any problems in sitting. Deformity and range of motion measurements are excluded from the standard HHS in order to allow remote completion.
  This assessment is recorded by a clinician onto the CRF via interview with the subject.
EQ-5D | 8 weeks, 12 weeks, 6 months and 12 months post-surgery
  The EuroQol EQ-5D is a standardized instrument for use as a measurement of health outcome. It consists of a descriptive system with 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) which are each assigned three levels (no problems, some problems, extreme problems) and a Visual Analogue Scale where subjects indicate a numerical value from 0-100 where 0 is the worst imaginable health state and 100 is the best imaginable health state.
  The EQ-5D is a patient reported outcome.
Log of opioid medication administered | Daily from day 1 post-surgery to discharge (estimated 2 weeks post-surgery)
  A daily assessment of opioid usage will be made including recording;
  • For each adminstration;
  * Drug
  * Dose
  * Route of administration
  * Time of administration

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Mitchell, MBChB FRCS, Principal Investigator — University Hospitals Bristol and Weston NHS Foundation Trust
Locations (5):
- United Kingdom (5):
  - Royal Devon and Exeter Hospital, Exeter
  - Gloucestershire Royal Hospital, Gloucester
  - Royal Liverpool University Hospital, Liverpool
  - Derriford Hospital, Plymouth
  - Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: No